CLINICAL TRIAL: NCT07287241
Title: Evaluation of Cardiac Function and Morphology in Individuals With Osteogenesis Imperfecta: Prospective Observational Study
Brief Title: Prospective Observational Cohort Study of Cardiac Structure and Function in Children and Adults With Osteogenesis Imperfecta
Acronym: OI Cardio
Status: Recruiting | Type: Observational
Sponsor: Istituto Ortopedico Rizzoli (Other)
Responsible Party: Sponsor
Other Study IDs: 665/2021/Oss/IOR
Record Dates: First submitted 2025-11-25; First posted 2025-12-17 (Actual); Last update posted 2025-12-17 (Actual); Status verified 2025-12

CONDITIONS: Osteogenesis Imperfecta (OI); Osteogenesis Imperfecta
Keywords: Osteogenesis Imperfecta; Bone Diseases; Musculoskeletal Diseases; Genetic Diseases; Observational Study
MeSH Terms: conditions — Osteogenesis Imperfecta; Bone Diseases; Musculoskeletal Diseases; Genetic Diseases, Inborn

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Osteogenesis Imperfecta patients
  Interventions: Other: Imaging evaluation, Echocardiography

INTERVENTIONS:
Other: Imaging evaluation, Echocardiography — Since this is an observational study, researchers collect general information from instrumental investigations and functional assessments carried out as part of normal clinical practice

SUMMARY:
This prospective observational investigation will examine the incidence and progression of cardiologic findings in individuals with OI across different age groups. Cardiopulmonary complications are recognized as major contributors to morbidity and mortality in adults with OI, although life expectancy has significantly improved in recent years due to medical advancements.

By systematically evaluating cardiovascular involvement in this population, the study aims to generate clinically relevant evidence to inform early cardiologic screening strategies and support the development of harmonized and targeted management approaches, ultimately improving clinical practice and the quality of life of individuals living with OI.

DETAILED DESCRIPTION:
Research on extra-skeletal manifestations, particularly those affecting the cardiovascular system, is still rather limited, despite this being one of the main causes of morbidity and mortality among these patients. Cardiovascular abnormalities can also be found in childhood, even in cases of mild Osteogenesis Imperfecta.

This observational prospective cohort study is to evaluate the presence and progression of structural and functional cardiac abnormalities in children and adults with Osteogenesis Imperfecta (OI).

Participants will undergo routine clinical and instrumental evaluations performed during standard follow-up visits at the study center, including:

* Clinical and genetic assessment
* Echocardio, electrocardiogram, and cardiology visit
* Radiographic evaluation
* Quality-of-life questionnaire (EQ-5D)

These assessments will be performed at baseline and periodically over a 60-month follow-up period to characterize cardiovascular involvement in OI and support early cardiologic screening strategies.

The Department of Rare Skeletal Disorders at Istituto Ortopedico Rizzoli, Bologna, Italy, has been a reference centre, and coordinating centre, of ERN BOND, the European Reference Network for rare BONe Diseases (https://ernbond.eu/), since its creation in 2017

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of OI according to the modified Sillence classification (Mortier et al., 2019)
* All subjects with OI who attend genetic consultations at the clinic affiliated with the Rare Skeletal Diseases Unit of the IRCCS Rizzoli Orthopaedic Institute (IOR)
* Willingness to undergo clinical and instrumental assessments at the IOR

Exclusion Criteria:

* Acute upper and/or lower respiratory tract infections at the time of assessment
* Cognitive impairment affecting cooperation and the performance of examinations

Ages: 5 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients affected by Osteogenesis Imperfecta
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2025-06-10 (Actual); Primary Completion 2031-12 (Estimated); Study Completion 2031-12 (Estimated)

PRIMARY OUTCOMES:
Cardiac abnormalities | From enrollment to the end of study at 60 months
  The incidence of structural and functional cardiac abnormalities in individuals with osteogenesis imperfecta.

CONTACTS AND LOCATIONS:
Locations (1):
- IRCCS Istituto Ortopedico Rizzoli, Bologna, Emilia-Romagna, Italy